CLINICAL TRIAL: NCT05146895
Title: Evaluation of Local Hyperthermia for the Treatment of Flat Warts After 4 Months: a Single-center, Single-blind, Randomized Controlled Trial
Brief Title: A Cohort Study of Hyperthermia and Imiquimod for the Treatment of Flat Warts
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Gao Xinghua, professor, First Hospital of China Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HH20190606
Record Dates: First submitted 2021-08-17; First posted 2021-12-07 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Human Papilloma Virus
Keywords: hyperthermia; human papillomavirus virus; flat warts
MeSH Terms: conditions — Hyperthermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local Hyperthermia at 44℃ for falt warts (Experimental): Local hyperthermia at 44℃ for 30 mins on one lesion region, at days of 1,2,3, 15, 16, 21 and 28.
  Interventions: Device: Local Hyperthermia at 44℃
- Imiquimod for Flat Warts (Active Comparator): Miquimod treatment: 3 times a week for 1 month
  Interventions: Drug: Imiquimod treatment

INTERVENTIONS:
Drug: Imiquimod treatment — As an control arm, for patients with flat warts
  Arms: Imiquimod for Flat Warts
Device: Local Hyperthermia at 44℃ — As an experimental arm, for patients with flat warts
  Arms: Local Hyperthermia at 44℃ for falt warts

SUMMARY:
flat warts are a superficial viral skin disease, extremely common in childhood.Treatment of warts is often difficult and involves different destructive procedures.Although several pharmacological and physical topical treatments are available (keratolytic agents, electrosurgery, cryotherapy, carbon dioxide laser), results are often unsatisfactory in terms of efficacy (frequent recurrence) and cosmetic outcome (scars, inflammatory reactions, transient or permanent hyper- or hypopigmentation).

Mild local Hyperthermia with a certain temperature range has been successfully used in the treatment of some diseases. It has been utilised in the treatment of some neoplasm, fungal and HPV infections. Investigators' study found that local hyperthermia at 44°C could cleared HPV in more than half of the patients with plantar warts. Investigators also note the fact that in patients with multiple lesions, the clearance of the target lesion is commonly followed by clearance of other distant lesions, a phenomenon suggesting that local hyperthermia could aid in establishing a specific immune response to eliminate HPV.So the purpose of the study is to evaluation local hyperthermia in the treatment of flat warts Appropriate control arms were designed for different conditions.

ELIGIBILITY:
Inclusion Criteria:

* 12-65 years old;
* diagnosis confirmed;
* signed informed consent

Exclusion Criteria:

* Pregnant woman;
* Local or systematic treatment within 3 months;
* Comorbidity of other severe gynecological inflammation,
* Infection, or tumor;
* Comorbidity of other serious illnesses;
* No guarantee of timely treatment and follow-up

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-10-20 (Actual); Primary Completion 2022-06-20 (Estimated); Study Completion 2022-06-20 (Estimated)

PRIMARY OUTCOMES:
clearance rates of HPV | 3 months after the last time of treatment
  to evaluate the clearance rates of all lesions in different treatment groups 3 month after treatment.

SECONDARY OUTCOMES:
effective rates of HPV | 3 months after the last time of treatment
  to evaluate the effective rates of all lesions in different treatment groups 3 month after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Hospital of China Medical University, Shenyang, China

IPD SHARING:
Plan to Share IPD: No